CLINICAL TRIAL: NCT05303506
Title: Prospective Study on the Effect of Different Risk Factors on the Growth Parameters of Thalassemic Patients in Assiut University Children Hospital (AUCH)
Brief Title: Study on the Effect of Different Risk Factors on the Growth Parameters of Thalassemic Patients in Assiut (AUCH)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Elmostafa Mohamed Hemida, mhemida92@gmail.com (resident physician of pediatrics), Assiut University
Other Study IDs: thalassemia in AUCH
Record Dates: First submitted 2021-11-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum ferritin and AST — observiational study

SUMMARY:
To assess the effect of different risk factors on the growth parameters of thalassemic patients in Assiut University children Hospital (AUCH) In order to help in decreasing the morbidity and mortality resulting from iron overload and improving the quality of life for thalassemic patient

DETAILED DESCRIPTION:
Thalassemia major is a heterogeneous disease presenting during infancy or early childhood. Although thalassemia is preventable by premarital counseling and prenatal testing, a large number of children are born with thalassemia, and curative treatment in the form of bone marrow or stem cell transplantation is not possible for the majority of these patients. Such patients need regular transfusions of packed red blood cells (PRBCs) Excess iron can potentially penetrate cells in the liver, heart, endocrine glands and other organs, Iron overload in the heart and liver is known to be a leading cause of morbidity and mortality among patients with transfusion-dependent b-thalassemia major Physical growth is affected in a large number of the patients with transfusion-dependent thalassemia. A study of patients aged 10-27 years with thalassemia major found short stature in 70% of the males and in 73% of the females, thalassemic patients are short, have low rate of growth and BMI and have either delayed or absent pubertal spurt, which is related to low hemoglobin and high ferritin levels and sub-optimal iron chelation therapy. (Najafipour, et al 2008 ).

Therefore, iron-chelating agents, such as deferoxamine, have been used since 1970 and has shown to be effective in chelating iron from the heart and liver, with preservation of heart function and reversal of hepatic fibrosis, respectively Recent advances in the medical management of regular blood transfusion and chelation therapy have allowed most of these patients to have improved survival well into adult life and improved quality of life in patients with severe b-thalassemia promote normal growth, allow normal physical activities, minimize transfusional iron accumulation, adequately suppress bone marrow activity and reduce cardiac overload due to chronic anemia .

Hemoglobin levels maintained at 9-10 g/dl are thought of as optimal , A higher target pre-transfusion hemoglobin level of 11-12 g/dl may be appropriate for patients with heart disease or other medical conditions There is a clear link between the overall iron burden and global toxicity; in patients with thalassemia the liver iron concentration correlates with the total body iron load Serum ferritin and liver iron concentration are widely used to detect iron overload, and the latter can be measured by magnetic resonance imaging (MRI), or liver biopsy, Evidence indicates that serum ferritin is not an accurate measure iron overload and that direct measurement of liver iron concentration via liver biopsy or MRI is more precise

ELIGIBILITY:
Inclusion Criteria:

* All children attending haematology unit in Assiut University Children Hospital with thalassemia treated by iron chelating agents and aged from one year to 16 years old.

Exclusion Criteria:

* Children not treated by chelating agents. Children with stem cell transplantation . Children with thalassemia minor or intermedia.

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: All children attending haematology unit in Assiut University Children Hospital with thalassemia treated by iron chelating agents and aged from one year to 16 years old.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-02 (Estimated); Primary Completion 2023-12-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Measuring the Effect of different risk factors on the Growth Parameters of Thalassemic Patients in Assiut University Children Hospital (AUCH) and how these risk factors affect the quality of life by measuring anthropocentric measures | 2 years
  Data of the patients will be collected from thalassemic patients in form of
  1. Personal history (Name, Age ,Sex)
  2. Therapeutic history (Age of diagnosis , Age of 1st chelator ,Chelator type , Chelator dose , Compliance to treatment )
  3. Growth parameters (Weight , Height,and mid arm circumference))
Decreasing the morbidity and mortality and improving the quality of life for thalassemic patient | 6 months
  At the end of the study there will be recommendations to help in decreasing the morbidity and mortality and improving the quality of life for thalassemic patient

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] . Pemde et al, publisher and licensee Dove Medical Press Ltd. This is an Open Access article which permits unrestricted noncommercial use, provided the original work is properly cited. Pediatric Health, Medicine and Therapeutics 2011:2 13-19
- [Background] Hoffbrand AV, Taher A, Cappellini MD. How I treat transfusional iron overload. Blood. 2012 Nov 1;120(18):3657-69. doi: 10.1182/blood-2012-05-370098. Epub 2012 Aug 23. PMID 22919029
- [Background] Rachmilewitz EA, Giardina PJ. How I treat thalassemia. Blood. 2011 Sep 29;118(13):3479-88. doi: 10.1182/blood-2010-08-300335. Epub 2011 Aug 2. PMID 21813448
- [Background] Najafipour F, Aliasgarzadeh A, Aghamohamadzadeh N, Bahrami A, Mobasri M, Niafar M, Khoshbaten M. A cross-sectional study of metabolic and endocrine complications in beta-thalassemia major. Ann Saudi Med. 2008 Sep-Oct;28(5):361-6. doi: 10.5144/0256-4947.2008.361. PMID 18779644
- [Background] Wood JC, Kang BP, Thompson A, Giardina P, Harmatz P, Glynos T, Paley C, Coates TD. The effect of deferasirox on cardiac iron in thalassemia major: impact of total body iron stores. Blood. 2010 Jul 29;116(4):537-43. doi: 10.1182/blood-2009-11-250308. Epub 2010 Apr 26. PMID 20421452
- [Background] Deugnier Y, Turlin B, Ropert M, Cappellini MD, Porter JB, Giannone V, Zhang Y, Griffel L, Brissot P. Improvement in liver pathology of patients with beta-thalassemia treated with deferasirox for at least 3 years. Gastroenterology. 2011 Oct;141(4):1202-11, 1211.e1-3. doi: 10.1053/j.gastro.2011.06.065. Epub 2011 Jul 7. PMID 21741344
- [Background] Cabantchik ZI, Breuer W, Zanninelli G, Cianciulli P. LPI-labile plasma iron in iron overload. Best Pract Res Clin Haematol. 2005 Jun;18(2):277-87. doi: 10.1016/j.beha.2004.10.003. PMID 15737890
- [Background] Borgna-Pignatti C. Surviving with thalassemia major: the Italian experience. Pediatr Hematol Oncol. 2007 Jan-Feb;24(1):75-8. doi: 10.1080/08880010601001461. No abstract available. PMID 17130117
- [Background] Wood JC, Enriquez C, Ghugre N, Tyzka JM, Carson S, Nelson MD, Coates TD. MRI R2 and R2* mapping accurately estimates hepatic iron concentration in transfusion-dependent thalassemia and sickle cell disease patients. Blood. 2005 Aug 15;106(4):1460-5. doi: 10.1182/blood-2004-10-3982. Epub 2005 Apr 28. PMID 15860670